CLINICAL TRIAL: NCT06352736
Title: Status of Disease Burden of Lower Urinary Tract Symptoms in Chinese Male Community
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qing Yuan, Professor, Chinese PLA General Hospital
Other Study IDs: LUTS2023
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Chinese community male population; Prevalence rate
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 5ml whole blood and 5ml urine per subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study, set up as a cross-sectional survey, seeks to delve into the disease burden and the demographic specifics of lower urinary tract symptoms (LUTS) among the male community in China. The investigators's main aim is to map out the overall and age-specific prevalence rates of LUTS within the Chinese male population. These insights are critical for understanding the public health dimensions of this condition. Moreover, the investigators plan to investigate several secondary aspects: the correlation of LUTS prevalence with factors like urbanization levels (rural vs. urban), geographical distribution, and lifestyle choices. Another significant focus will involve examining the treatment landscape for LUTS, looking at the portion of sufferers receiving treatment, the diversity in treatment durations, and the types of treatments employed (medication vs. surgery). This comprehensive analysis is intended to shed light on the prevailing management strategies for LUTS in China. The study is scheduled to unfold over 36 months and will comprise three pivotal phases: initial preparations, recruitment of subjects and collection of data, followed by the analysis of data and compilation of reports. The investigators will employ a range of methods such as questionnaires, physical exams, laboratory tests, imaging, and other medical evaluations to amass extensive data. This will allow the investigators to evaluate the prevalence of LUTS across various age groups among men and address the current gaps in epidemiological understanding.

DETAILED DESCRIPTION:
Divide the country into 7 geographical regions and stratify them according to urban and rural areas. Based on the size of the male population over 40 years old in the seventh National Census, employ a multi-stage proportional-to-size (PPS) sampling method. The sampling process is divided into six stages. In the first stage, use provincial-level administrative units as sampling units. Based on population size, use the PPS method to select 2 provincial-level administrative units from each region, totaling 14. In the second stage of sampling, use prefecture-level cities in each province as sampling units. The capital cities are directly sampled; based on population size, use the PPS method to select 1 other prefecture-level city from each province. In the third stage of sampling, use urban districts and counties (including county-level cities) in prefecture-level cities/direct-controlled municipalities as sampling units. Use the PPS method to select 2 urban districts and 2 counties in each prefecture-level city, and 4 urban districts and 4 counties in each direct-controlled municipality. In the fourth stage of sampling, use streets in urban districts and towns/townships in counties as sampling units. Use simple random sampling to select 1 street from each urban district and 1 town/township from each county. In the fifth stage of sampling, use communities in streets and villages in towns/townships as sampling units. Use simple random sampling to select 2 communities from each street and 2 villages from each town/township. In the sixth stage of sampling, stratify males over 40 years old in each community/village by age groups (40-49 years,50-59 years,60-69 years,70 years and above). Number individuals of each age group and randomly sample individuals. This survey includes four parts: questionnaire survey, physical examination, laboratory tests, imaging and other examinations. The questionnaire is conducted face-to-face by trained interviewers.

ELIGIBILITY:
Inclusion Criteria:

1. Mainland China, aged 40 or older, male, in 31 provincial-level administrative regions.
2. Have resided for a total of 6 months or more in the survey county (district) in the past 12 months.
3. Normal communication, cooperation during physical examination, and good cognitive ability.
4. Willing to participate in and cooperate with this study, and sign the informed consent form.

Exclusion Criteria:

1. Closed communities, such as armed forces and nursing homes.
2. Individuals with mental illnesses or other conditions that prevent cooperation.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 12567 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score(IPSS) | DAY 1
  A questionnaire to assess the condition of the prostate, report by score.The minimum value is 0, the maximum is 35, and the larger the score, the more severe the symptoms.
Overactive Bladder Syndrome Score(OABSS) | Day 1
  A questionnaire to assess the condition of overactive bladder, report by score.The minimum value is 0, the maximum is 15, and the larger the score, the more severe the symptoms.The minimum value is 0, the maximum is 15, and the larger the score, the more severe the symptoms.
International Consultation on Incontinence Questionnaire - Short Form(ICIQ-SF) | Day 1
  Detection through urinary flow rate meter, report by score.The minimum value is 0, the maximum is 11, and the larger the score, the more severe the symptoms
Quality of Life Score（QOL） | Day 1
  t was used to assess the impact of lower urinary tract symptoms on quality of life, with a minimum score of 0 and a maximum score of 6. The smaller the score, the higher the quality of life.

SECONDARY OUTCOMES:
Prostatic volume | Day 1
  By transabdominal ultrasound, Prostatic volume (ml)= Lateral diameter of prostate(cm)* Anterior and posterior prostatic diameter(cm) * Diameter superior and inferior prostatic (cm) *0.52
Maximum urinary flow rate | Day 1
  Detection through urinary flow rate meter （ml/min)
Residual urine | Day 1
  By transabdominal ultrasound (ml)
free prostatic specific antigen(fPSA) | Day 1
  ng/ml
total prostatic specific antigen(tPSA) | Day 1
  ng/ml
fPSA/ tPSA | Day 1
  fPSA/ tPSA, Ratio of the two

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The data involves a large amount of personal information and privacy of the population, and the informed consent promises the confidentiality of personal data.

REFERENCES:
- [Background] Lerner LB, McVary KT, Barry MJ, Bixler BR, Dahm P, Das AK, Gandhi MC, Kaplan SA, Kohler TS, Martin L, Parsons JK, Roehrborn CG, Stoffel JT, Welliver C, Wilt TJ. Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA GUIDELINE PART I-Initial Work-up and Medical Management. J Urol. 2021 Oct;206(4):806-817. doi: 10.1097/JU.0000000000002183. Epub 2021 Aug 13. PMID 34384237
- [Background] Nambiar AK, Arlandis S, Bo K, Cobussen-Boekhorst H, Costantini E, de Heide M, Farag F, Groen J, Karavitakis M, Lapitan MC, Manso M, Arteaga SM, Riogh ANA, O'Connor E, Omar MI, Peyronnet B, Phe V, Sakalis VI, Sihra N, Tzelves L, van Poelgeest-Pomfret ML, van den Bos TWL, van der Vaart H, Harding CK. European Association of Urology Guidelines on the Diagnosis and Management of Female Non-neurogenic Lower Urinary Tract Symptoms. Part 1: Diagnostics, Overactive Bladder, Stress Urinary Incontinence, and Mixed Urinary Incontinence. Eur Urol. 2022 Jul;82(1):49-59. doi: 10.1016/j.eururo.2022.01.045. Epub 2022 Feb 23. PMID 35216856
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Chapple C, Castro-Diaz D, Chuang YC, Lee KS, Liao L, Liu SP, Wang J, Yoo TK, Chu R, Sumarsono B. Prevalence of Lower Urinary Tract Symptoms in China, Taiwan, and South Korea: Results from a Cross-Sectional, Population-Based Study. Adv Ther. 2017 Aug;34(8):1953-1965. doi: 10.1007/s12325-017-0577-9. Epub 2017 Jul 7. PMID 28687936
- [Background] Chow PM, Chuang YC, Hsu KCP, Shen YC, Hsieh AW, Liu SP. Impacts of nocturia on quality of life, mental health, work limitation, and health care seeking in China, Taiwan and South Korea (LUTS Asia): Results from a cross-sectional, population-based study. J Formos Med Assoc. 2022 Jan;121(1 Pt 2):285-293. doi: 10.1016/j.jfma.2021.04.005. Epub 2021 May 4. PMID 33958270
- [Background] Zhang W, Cao G, Sun Y, Wu F, Wang Q, Xu T, Hu H, Xu K. Depressive symptoms in individuals diagnosed with lower urinary tract symptoms suggestive of benign prostatic hyperplasia (LUTS/BPH) in middle-aged and older Chinese individuals: Results from the China Health and Retirement Longitudinal Study. J Affect Disord. 2022 Jan 1;296:660-666. doi: 10.1016/j.jad.2021.09.045. Epub 2021 Sep 20. PMID 34565588